CLINICAL TRIAL: NCT06431009
Title: The Danish Region Midt Schizophrenia (RMS) Cohort: Representative Cohort of Patients With a First-episode Schizophrenia Spectrum Disorder With Long-term Follow-up
Brief Title: The Danish Region Midt Schizophrenia Cohort
Acronym: RMS
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-001
Record Dates: First submitted 2024-02-23; First posted 2024-05-28 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotics; Adverse Childhood Experiences (ACE); Immune system
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Schizophrenia: Patients with a SSD (ICD-10: F20-29) aged ≥15 years.
  Interventions: Other: Treatment-as-usual
- Ultra High Risk: Patients at UHR (ICD: 1*.5) aged ≥15 years.
  Interventions: Other: Treatment-as-usual

INTERVENTIONS:
Other: Treatment-as-usual — Patients will be treated and followed according to normal clinical treatment guidelines at the local psychiatric hospitals, which will not be affected by participation in the RMS cohort.

SUMMARY:
The objective of this study is to recruit patients at the first diagnosis with a schizophrenia spectrum disorder (SSD) and ultra-high risk patients (UHR), defined as patients with drug abuse and psychotic symptoms indicating a risk for developing schizophrenia. Thereby, the investigators aim to establish a large representative cohort of patients with a first-episode SSD or patients at UHR, enabling investigations of the etiology and long-term prognosis of SSDs. The primary aim is to learn more about the importance of adverse childhood experiences (ACEs) and the immune system in the etiology and course of schizophrenia. Patients will be followed with planned visits after 1, 2, 3, 12 and 24 months including online questionnaires after 2, 6, 10 and 26 weeks. There will be the possibility to contact patients again for subsequent follow-up visits.

DETAILED DESCRIPTION:
Study design: Cohort study with pre-defined longitudinal follow-up visits. Patients: Patients with a SSD (ICD-10: F20-29) or patients at UHR (ICD: 1*.5) aged ≥15 years.

Sample size: Within the Central Denmark Region (CDR), approximately 700 patients are each year diagnosed with a SSD and 100 with UHR. The investigators will establish recruitment at all psychiatric hospitals in the CDR between January 2024 until June 2025. Our aim is to establish continued recruitment of 100-150 patients/year. Hence, the investigators expect to recruit 300-350 patients during the period 2024-2026.

Procedures: Patients will be included within three months of the first SSD or UHR diagnosis at one of the psychiatric hospitals in the CDR. Before inclusion, an interview with the Schedules for Clinical Assessment in Neuropsychiatry (SCAN) interview will validate the diagnosis. At baseline and follow-up visits (details in the full protocol and Table 1), patients will be rated by use of the 6-item Positive and Negative Syndrome Scale (PANSS-6), the Clinical Global Impression Severity Scale (CGI-S), the Global Assessment of Functioning Scale (GAF), the Schizophrenia Quality of Life Scale (SQLS), Alcohol Use Disorders Identification Test (AUDIT), Drug Use Disorders Identification Test (DUDIT), Fagerström Test for Nicotine Dependence (FTND), Major Depression Inventory (MDI), the Aarhus Side effect Assessment Questionnaire (ASAQ), the "Udvalg for Kliniske Undersøgelser" side effect scale (UKU), and the Calgary Depression Scale for Schizophrenia (CDSS). Furthermore, patients will fill out the self-reported WHO Adverse Childhood Experience International Questionnaire (ACE-IQ) and the Insomnia Severity Index (ISI), the Epsworth Sleepiness Scale (ESS), and the Pittsburgh Sleep Quality Index (PSQI) to measure sleep. The Matrics Consensus Cognitive Battery (MCCB), which consists of 10 cognitive tests, will measure cognition. To measure consciousness, patients will fill out the Perceived Stress Scale (PSS), Toronto Alexithymia Scale (TAS-20), and Metacognition Superiority illusion. During the first three months, participants will wear an actigraph to have a proxy measure of activity and sleep. Blood sampling will be performed at baseline and after 3, 12 and 24 months to measure markers of inflammation and to enable genetic and epigenetic analyses. Heart rate, blood pressure, height, body weight, waist and hip circumference will be recorded. Patients will be treated according to clinical indication, i.e., they will receive routine clinical care at the local psychiatric hospital and participation in this study will not affect the treatment. Patients can be included in this study independent of whether they are treated with psychotropic drugs or not.

Follow-up: Patients will be treated and followed according to normal clinical treatment guidelines at the local psychiatric hospitals, which will not be affected by participation in the RMS cohort. Patients will have follow-up visits for the RMS study after 1, 2, 3, 12 and 24 months after the individual inclusion date and fill out online questionnaires after 2, 6, 10, and 26 weeks.

Endpoints: The primary endpoint is the correlation between ACEs and inflammatory markers measured at baseline with the change on PANSS-6 from baseline to follow-up visits. Key secondary endpoints include changes in genetic, epigenetics, cognition, PSQI and ISI. Additional secondary endpoints include changes in ASAQ, UKU, SQLS, CDSS, GAF, CGI-S, body weight, hip and waist circumference, blood pressure, and heart rate. For patients enrolled in the study, all endpoints will initially be collected and several repeated during the study duration.

Safety: Patients will follow treatment-as-usual at their local hospital, with the clinicians from the local hospital being responsible for safety monitoring according to local treatment guidelines. Blood sample results will be obtained from the patient's medical record (MidtEPJ) at the study visits to monitor biochemical safety parameters for medical treatment. Between follow-up visits for the RMS cohort, patients will follow guideline-based safety monitoring at the local psychiatric hospital.

Study duration: Continuous. The investigators aim to establish continuous recruitment and that all patients with a first-episode SSD or UHR diagnosis fulfilling inclusion criteria will be offered participation in the RMS Cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥15 years
2. Diagnosed within the previous 3 months with first-episode SSD (ICD-10: F20-29) or UHR (ICD-10: F1X.5)
3. Able to give informed oral and written consent.

Exclusion Criteria:

1. Any coercive measure including patients in forensic psychiatry
2. In a clinical condition where the treating clinician evaluates that the patient is not able to attend the research study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient aged ≥15 years diagnosed with first-episode SSD or UHR diagnosis and without any coercive measure at the time of inclusion will be relevant for inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse childhood experiences (ACEs) | from baseline to follow-up visits after 52 and 104 weeks.
  The primary endpoint is the correlation between adverse childhood experiences (ACEs, from 0 to 13 ACEs measured via the World Health Organization (WHO) ACE-IQ), reported at baseline, with the change on the 6-item positive and negative symptom scale (PANSS-6, minimum score=0, maximum score=30), with higher PANSS-6 scores indicating greater symptom severity

SECONDARY OUTCOMES:
Cognition | from baseline to follow-up visits after 52 and 104 weeks.
  Changes in cognition, measured via matrics consensus cognitive battery (MCCB, presenting T-scores (minimum=0, maximum=60) for 7 different cognitive domains) with higher scores indicating better cognitive functioning
Sleep | from baseline to follow-up visits after 52 and 104 weeks.
  Changes in sleep quality (measured via Pittsburgh Sleep Quality Index (PSQI, minimum score=0, maximum score=39) and Insomnia Severity Index (ISI, minimum score=0, maximum score=28), with both measures indicating worse sleep quality depending on higher scores on the scales)
Quality-of-life | from baseline to follow-up visits after 52 and 104 weeks.
  Changes in quality-of-life (measuring psychosocial quality-of-life, energy+motivation, and symptoms+side effects via the Schizophrenia Quality of Life Scale (SQLS, minimum score=0, maximum score=30), with higher scores indicating worse quality-of-life)
Level of functioning | from baseline to follow-up visits after 52 and 104 weeks.
  Changes in level of functioning, (measured via the Global Assessment of Functioning (GAF), with higher scores on a scale from 0 to 100 indicating better functioning)

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Aarhus University Hospital Psychiatry, Aarhus
  - Psychiatric Hospital Gødstrup, Herning
  - Psychiatric Hospital Horsens, Horsens
  - Psychiatric Hospital Randers, Randers
  - Psychiatric Hospital Midt, Silkeborg

IPD SHARING:
Plan to Share IPD: No